CLINICAL TRIAL: NCT02754999
Title: An Open-label Phase 1 Safety Study of SANGUINATE™ Infusion in Patients With Acute Severe Anemia Who Are Unable to Receive Red Blood Cell Transfusion
Brief Title: A Phase 1 Safety Study of SANGUINATE™ In Patients With Acute Severe Anemia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGHY-001
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Acute Anemia
MeSH Terms: interventions — PEGylated carboxyhemoglobin bovine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SANGUINATE™ (Experimental): As Needed Dosing of SANGUINATE
  Interventions: Drug: SANGUINATE™

INTERVENTIONS:
Drug: SANGUINATE™ — As needed (PRN) infusions of 500 mL of SANGUINATE
  Other Names: pegylated carboxyhemoglobin bovine

SUMMARY:
In this open-label study, eligible and consenting adult patients admitted to the hospital for critical care that have acute severe anemia, defined as a blood hemoglobin level ≤ 5 g/dL, but who are unwilling or unable to receive red blood cell (RBC) transfusion, will receive one or more infusions of SANGUINATE as are deemed necessary by the Investigator for survival of the acute anemic episode.

DETAILED DESCRIPTION:
Data collection for each patient during the in-patient portion of the study will be required for up to a maximum of 14 days while under critical care, with additional collection of safety-related findings at 7 days and 14 days after the last infusion of SANGUINATE. Each patient will thus have up to 28 days participation in the trial.

A minimum of 100 subjects are to be enrolled and to receive at least one infusion of SANGUINATE, with 14-day follow-up after the last infusion.

Because of the life-threatening effects of severe anemia, it is expected that all patients in this trial will receive care within a critical care facility (may be called intensive care or some similar name), wherein all patients will have real-time monitoring of vital signs and ECG (e.g., by telemetry) before, during, and after all study drug infusions.

ELIGIBILITY:
Inclusion Criteria:

1. The patient would otherwise receive RBC transfusion for treatment of severe anemia but cannot (hemolytic/allosensitized or no compatible blood) or will not (religious/personal objection) receive RBCs
2. Hemoglobin ≤ 5 g/dL, or hemoglobin ≤ 7 g/dL following a decline of ≥ 5 g/dL over less than 7 days
3. Age ≥ 18 years
4. Receiving or willing to receive supplemental iron therapy (unless contraindicated)
5. Receiving or willing to receive erythropoiesis-stimulating agent (EPO) therapy
6. Patient or legally authorized representative provided consent to participate
7. Investigator determination that the patient is an appropriate candidate for study enrollment

Exclusion Criteria:

1. Hemoglobin ≤ 2 g/dL
2. Presence of severe trauma (e.g., Injury Severity Score (ISS)/New Injury Severity Score (NISS) Score ≥ 25)
3. Unable to provide sufficient blood sample volume for screening assessments; or
4. Pregnant; or
5. Investigator determination that the patient is not an appropriate candidate for study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events within 24-hours of each SANGUINATE infusion | 24 Hours
  Composite endpoint defined by changes in vital signs, electrocardiographic, biochemical, hematological, and urinalysis, death and other reported adverse events

SECONDARY OUTCOMES:
Percentage of patients who survive the acute episode of severe anemia | 14 Days
Percentage of patients who recover from hypoxia-induced abnormal end-organ function | 14 Days
Percentage of patients who improved with their hemodynamic status | 14 Days
Percentage of patients who discontinue inotrope therapy | 14 Days
Percentage of patients who discontinue respiratory support/therapy | 14 Days
Number of serious adverse events following the start of SANGUINATE infusions through the final visit (up to 28 days) | 28 Days
  Composite endpoint defined by changes in vital signs, electrocardiographic, biochemical, hematological, and urinalysis, death and other reported serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Abe Abuchowski, PhD, Study Director — Prolong Pharamceuticals
Locations (32):
- United States (32):
  - Brookwood Princeton Baptist, Birmingham, Alabama
  - Yavapai Regional Medical Center, Prescott, Arizona
  - Kaiser Permanente, Baldwin Park, California
  - City of Hope, Duarte, California
  - Antelope Valley Hospital, Lancaster, California
  - Loma Linda Medical Center, Loma Linda, California
  - Providence Holy Cross Hospital, Mission Hills, California
  - Medstar Georgetown University Hosiptal, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Wellstar Atlanta Medical Centre, Marietta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Detroit Medical Center Harper Univesity Hospital, Detroit, Michigan
  - Englewood Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Barnabas, Livingston, New Jersey
  - Northwell - North Shore University Hospital, Lake Success, New York
  - Mt. Sinai /Recanati/Miller Transplantation Institute, Icahn, New York, New York
  - Presbyterian Hospital Novant Health, Charlotte, North Carolina
  - Abington University, Abington, Pennsylvania
  - Hahnemann University Hospital (Rittenhouse), Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Bon Secour St Francis Cancer Center, Greenville, South Carolina
  - University of Texas Medical Center (El Paso), El Paso, Texas
  - Houston Methodist Hospital, Houston, Texas
  - St. Lukes, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No